CLINICAL TRIAL: NCT00433823
Title: A Multicenter, Open Labeled, Cross-Over Designed Prospective Study Evaluating the Effects of Lipid Lowering Treatment on Steroid Synthesis
Brief Title: A Study Evaluating the Effects of Lipid Lowering Treatment on Steroid Synthesis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Abant Izzet Baysal University (Other)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: MK-19
Record Dates: First submitted 2007-02-07; First posted 2007-02-12 (Estimated); Last update posted 2007-02-12 (Estimated); Status verified 2007-02

CONDITIONS: Coronary Heart Disease; Diabetes Mellitus; Non-Coronary Atherosclerotic Disease; Hypercholesterolemia
Keywords: Very low level of LDL; Steroid hormones; Atorvastatin; Ezetimibe; Lipoprotein-a
MeSH Terms: conditions — Coronary Disease; Diabetes Mellitus; Hypercholesterolemia | interventions — liptruzet

INTERVENTIONS:
Drug: Atorvastatin, Ezetimibe

SUMMARY:
Cholesterol is the precursor of glucocorticoids, mineralocorticoids and sex steroids. Both adrenal and non-adrenal (ovarian + testicular) all steroid hormones are primarily synthesized using the LDL-cholesterol in the circulation. Additionally there is 'de novo' cholesterol synthesis in both the adrenals and gonads controlled by the HMG-CoA reductase enzyme. A third pathway is the use of circulatory HDL-cholesterol by the adrenal and gonadal tissues for the synthesis of steroids. Since statins both decrease circulatory LDL and inhibit de novo cholesterol synthesis, they are likely to affect the synthesis of steroid hormones. In this study we aim to investigate the effects of lowering LDL levels below 70 mg/dL on steroid hormone synthesis.

DETAILED DESCRIPTION:
Today atherosclerotic diseases are among the most important causes of death in the world. Epidemiological, clinical, genetic, experimental and pathological studies have clearly shown the role of lipoproteins in atherosclerosis. LDL is the major atherogenic lipoprotein and has been defined as the primary target of lipid lowering treatment by NCEP. Although the level of LDL, the primary target in the treatment of dyslipidemia, has been set as below 100mg/dl in coronary heart diseases (CHD) and CHD risk equivalents, this level has been pulled down to below 70mg/dl for the group defined as very high risk group by the ATP (Adult Treatment Panel) guide that has been updated following the new clinical studies. As we already know, cholesterol is the precursor of glucocorticoids, mineralocorticoids and sex steroids, besides being a structural component of the cell membrane. Both adrenal and non-adrenal (ovarian+testicular) all steroid hormones are primarily synthesized using the LDL-cholesterol in the circulation. In addition to this, there is 'de novo' cholesterol synthesis in both the adrenals and gonads controlled by the HMG-CoA reductase enzyme. A third pathway, which under normal circumstances has little contribution as compared to the first two, is the use of circulatory HDL-cholesterol by the adrenal and gonadal tissues for the synthesis of steroids. Our knowledge on extremely lowered LDL levels is quite limited. However, since statins both decrease circulatory LDL and inhibit de novo cholesterol synthesis, they are likely to affect the synthesis of steroid hormones.

ELIGIBILITY:
Inclusion Criteria:

* Patients in the very high risk group according to the ATPIII guide.

Exclusion Criteria:

* Patients having a major disease involving hepatic, gastrointestinal and endocrinologic diseases other than diabetes.
* Patients having a known muscle disease
* Pregnancy, breast-feeding
* Patients having a history of allergy to statins or ezetimibe
* Nephropathic patients

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2007-01; Study Completion 2008-01

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Kanat, MD, Principal Investigator — Abant Izzet Baysal University, Bolu Izzet Baysal School of Medicine
Locations (1):
- Bolu Izzet Baysal School of Medicine, Bolu, Turkey (Türkiye)